CLINICAL TRIAL: NCT02546180
Title: Improving Patient Understanding of the Surgical Hospital Experience: Use of YouTube Video Playlist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mary O'Connor, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB # 14-000084
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Anxiety
Keywords: Patient education; Preoperative anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- YouTube Video Viewers (Experimental): Subjects in this arm were randomized to viewing YouTube videos.
  Interventions: Other: Viewing YouTube videos
- Standard Education (Active Comparator): Subjects in this arm were randomized to standard preoperative education.
  Interventions: Other: Standard preoperative education

INTERVENTIONS:
Other: Viewing YouTube videos — The on-line patient education program will highlight postoperative care.
  Arms: YouTube Video Viewers
Other: Standard preoperative education — Standard preoperative education will be provided by the surgeon, physician extender and paramedical staff in the clinic.
  Arms: Standard Education

SUMMARY:
This prospective randomized pilot clinical trial studied the effect on preoperative anxiety of watching a series of YouTube videos designed to create a virtual hospital experience for patients undergoing primary total hip and knee arthroplasty as compared to routine preoperative education.

Hypothesis: Preoperative anxiety related to hip and knee replacement surgeries can be reduced by patient exposure to a virtual hospital inpatient experience delivered by a series of YouTube videos.

DETAILED DESCRIPTION:
As high patient anxiety prior to surgery has been linked to more severe and persistent pain after joint replacement surgery, the Orthopedic Surgery Department at Mayo Clinic in Florida created a playlist of 16 YouTube videos aimed at creating a virtual hospital experience for primary total hip and knee joint replacement patients. A pilot study was then performed to evaluate the potential impact of viewing this playlist on preoperative anxiety.

Methods: Each patient completed a Generalized Anxiety Disorder Score (GAD) assessment at the time of the routine preoperative clinic visit and were then randomized based on their gender, type of surgery, and initial GAD score to either the control group of standard education (education at face-to-face clinical visits as well as printed educational materials) or the treatment group of standard education plus access to the YouTube playlist. On the morning of the patient's surgery the same survey was repeated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary total hip or total knee arthroplasty at Mayo Clinic in Florida
* Patients must be able to give consent to the study
* Patients must agree to watch the videos prior to scheduled surgery
* Patients must agree to complete the questionnaire in the office and again prior to surgery on the day of surgery

Exclusion Criteria:

* No internet access at home
* Visual or auditory conditions which limit a patient's ability to view the You Tube videos at home

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Generalized Anxiety Disorder (GAD) Score | Baseline, approximately 2-3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary O'Connor, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- [Derived] O'Connor MI, Brennan K, Kazmerchak S, Pratt J. YouTube Videos to Create a "Virtual Hospital Experience" for Hip and Knee Replacement Patients to Decrease Preoperative Anxiety: A Randomized Trial. Interact J Med Res. 2016 Apr 18;5(2):e10. doi: 10.2196/ijmr.4295. PMID 27091674